CLINICAL TRIAL: NCT03918174
Title: Efficacy of Treatment After Distal Radius Fractures Using Dart-throwing Motion
Brief Title: Implementation of the Dart-throwing Motion Plane in Hand Therapy After Distal Radius Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-15-2085-YY-CTIL
Record Dates: First submitted 2019-04-01; First posted 2019-04-17 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Distal Radius Fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Intervention Model Description: After enrollment, subjects were randomly divided into the research group and into the control group. Both groups went through the same intake evaluation. On completion of the intervention, both groups were reevaluated and filled out a satisfaction questionnaire.
  The research group alone filled out the Quebec User Evaluation of Satisfaction with assistive Technology (QUEST) questionnaire, to measure the level of satisfaction attribute to assistive technologies, e.g., the innovative dart splint they exercised with.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dart Splint orthosis (Experimental): The Dart-Splint orthosis allows oblique wrist motion along the Dart Throwing Motion (DTM) plane, thus inhibiting movement of the healing structures following surgery around the distal radius. This is a hinged orthosis that permits selective midcarpal mobilization along the plane of the DTM is a novel orthotic device that was developed in order to facilitate protected midcarpal motion.
  Interventions: Device: Dart splint orthosis
- The conventional treatment (Experimental): The control group activated the wrist mostly in the sagittal plane. This group was instructed to perform at home active wrist motion similar to that practiced during the supervised therapy sessions. The prescribed instructions were similar to the exercises performed during the sessions.
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Device: Dart splint orthosis — The Dart Splint orthosis was fitted to the subjects in the research group on their first evaluation session. They received oral and written instructions regarding the donning and manner of exercise. Specifically, they were instructed to use the Dart splint orthosis at home. For each 10-minute exercise session, they were asked to perform 5 minutes of radial-extension under resistance and then 5 minutes ulnar-flexion under resistance. In addition, this group was required to fill in a chart at the end of each practice session (morning, noon and evening), throughout the intervention period.
  Other Names: Conventional treatment
  Arms: Dart Splint orthosis
Other: Conventional treatment — The control group activated the wrist mostly in the sagittal plane. This group was instructed to perform at home active wrist motion similar to that practiced during the supervised therapy sessions. The prescribed instructions were similar to the exercises performed during the sessions. Specifically, they were instructed to exercise at home for 10-minute in each session, three times a day (morning, noon and evening), throughout the intervention period.
  Arms: The conventional treatment

SUMMARY:
Rehabilitation following wrist fractures often includes exercising flexion-extension. However, during daily functions, our wrist moves through an oblique plane, named the Dart Throwing Motion (DTM) plane. This plane might be a more stable plane in cases of wrist injuries, since the proximal carpal row remains relatively immobile. However, rehabilitation programs that incorporate exercising in the DTM plane have yet to be explored.

The researchers aimed to evaluate the rehabilitation outcomes following treatment in the DTM plane compared with outcomes following treatment in the sagittal plane after Distal Radius Fracture (DRFs).

Twenty four subjects following internal fixation of DRFs were randomly assigned into a research group . The range of motion, pain levels and functional tests were measured before and after an intervention of 12 treatment sessions. The control group activated the wrist in the sagittal plane while the research group activated the wrist in the DTM plane, via a DTM orthosis.

DETAILED DESCRIPTION:
Twenty four subjects were recruited after Open Reduction Internal Fixation (ORIF) of DRFs. Inclusion criteria were: individuals aged 18 to 65 years. Individuals with previous orthopedic or neurological impairments of the upper limb or a cognitive impairment were excluded from the study. Subjects were enrolled from the department of hand surgery at the Sheba medical center.

Each subject read and signed an informed consent form pretrial. Each subject went through an intake session documenting personal information, upper limb ROM, pain levels and functional tests recorded by a certified occupational therapist (OT), hand therapist. The Sagittal group activated the wrist mostly in the sagittal plane while the research group activated the wrist also in the DTM plane, via the Modified Dart Splint (MDS).

All of the subjects in both groups received 12 therapy sessions, 30 minutes each one, 2-3 times a week, during 6-8 weeks following the removal of the cast. Certified hand therapists used several different treatment techniques during the sessions, to achieve the primary goals of edema control, increased Range of Motion (ROM), and decreased stiffness. Compressive wrap with retrograde massage, scar management, soft-tissue mobilization, joint mobilization, active motion and ROM exercises were practice patterns used in this study for all subjects, regardless their group. Both groups were instructed to exercise at home, 3 times a day, 10 minutes per exercise session. The MDS was fitted to the subjects in the DTM group on their first evaluation session. They received oral and written instructions regarding the donning and manner of exercise. Specifically, they were instructed to use the MDS at home. For each 10-minute exercise session, they were asked to perform 5 minutes of radial-extension under resistance and then 5 minutes ulnar-flexion under resistance. In addition, this group was required to fill in a chart at the end of each practice session (morning, noon and evening), throughout the intervention period. The researcher performed weekly phone calls to remind the DTM group to fill these out. The Sagittal group was instructed to perform at home active wrist motion similar to that practiced during the supervised therapy sessions. The prescribed instructions were similar to the exercises performed during the sessions.

At the completion of the treatment, the subjects were reexamined by the same evaluator that performed the baseline evaluation.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years old
* Went through open reduction internal fixation of distal radius fracture.

Exclusion Criteria:

* Individuals with previous orthopedic impairments of the upper limb.
* Individuals with neurological impairments of the upper limb.
* Individuals with a cognitive impairment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-11-15 (Actual); Primary Completion 2018-10-14 (Actual); Study Completion 2019-03-17 (Actual)

PRIMARY OUTCOMES:
A personal questionnaire | baseline
  6 questions regarding personal information (age, sex, family status, profession, hand dominance, and injured hand).
A house hold work and sport activity questionnaire | baseline
  10 questions regarding house hold activities (heavy housing and light housing) and sport activities (athletics, spinning, cycling, ball, racket, weights, swimming) were ranked on a Likert scale from 1-4 according to the daily, weekly or monthly amount of time put in to them.
Change in the forearm and wrist range of motion | Change from baseline forearm and wrist range of motion at two months
  The elbow and wrist active range of motions were measured during pro-supination, flexion-extension, radio-ulnar deviation. Additionally, the DTM plane angle of the wrist was measured according to Bugden's (Bugden, B. (2013). A proposed method of goniometric measurement of the dart-throwers motion. Journal of Hand Therapy, 26(1), 77-80. https://doi.org/10.1016/j.jht.2012.08.003)
Change in reported pain and function on The Patient-Rated Wrist Evaluation (PRWE) questionnaire. | Change from baseline pain and function at two months
  The PRWE is a 15-item questionnaire designed to measure wrist pain and disability in ADL (activities of daily living).
  The PRWE allows patients to rate their levels of wrist pain and disability from 0 to 10, and consists of 2 subscales:
  Pain subscale: contains 5 items each of which is further rated from 1-10. The maximum score in this section is 50 and minimum 0.
  Function subscale: contains total 10 items which are further divided into 2 sections i.e specific activities (having 6 items) and usual activities (having 4 items). The maximum score in this section is 50 and minimum 0.
Change in hand function on The Jebsen-Taylor Hand Function Test (JHFT) | Change from baseline hand function at two months
  The Jebsen-Taylor Hand Function Test (JHFT) was carried out to assess fine motor skills, weighted and non-weighted hand function activities during performance of ADLs and the effectiveness of treatment for hand conditions. Seven subsets of the test represent a broad spectrum of hand function, which includes writing, turning over 3x5 inch cards (to simulate page turning), picking up small common objects, simulated feeding, stacking checkers, picking up large light objects, and picking up large heavy objects. To evaluate patient performance, each subset is timed and can be compared to the established norms
Grip strength | Following the intervention at two months
  The Jamar hand dynamometer was used to measure grip strength. Grip strength was measured with the elbow flexed at 90° and the forearm in neutral rotation. A single measure of grip strength was performed during assessment. The second handle position of the dynamometer was used throughout testing.
Pinch strength | Following the intervention at two months
  The B&L engineering pinch gauge pinch meter was used to measure the three pinch strength outcomes: Lateral pinch, Tripod pinch and tip to tip pinch.
Satisfaction from the self-training | Following the intervention at two months
  Satisfaction from the self-training home exercises was rated using a 5-point Likert scale (1- Not satisfied to 5- Extremely satisfied) for 10 statements re self-training home exercises.
Quebec User Evaluation of Satisfaction with assistive Technology (QUEST) questionnaire | Following the intervention at two months
  The Quebec User Evaluation of Satisfaction with assistive Technology (QUEST) questionnaire, measured the level of satisfaction attributed to assistive technologies, i.e., the DTM orthosis (for the research group only). This questionnaire contained 27 variables which were scored in terms of perceived importance and satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Sigal Portnoy, PhD, Study Chair — Tel Aviv University

IPD SHARING:
Plan to Share IPD: No
Only statistical outcome measure are to be shared with other researchers.

DOCUMENTS (2):
  • Study Protocol (2015-05-11): https://cdn.clinicaltrials.gov/large-docs/74/NCT03918174/Prot_000.pdf
  • Statistical Analysis Plan (2015-05-11): https://cdn.clinicaltrials.gov/large-docs/74/NCT03918174/SAP_001.pdf